CLINICAL TRIAL: NCT03941938
Title: Prevention of Anastomotic Leak in Colorectal Surgery by Glue Reinforcement. A Prospective Randomized Trial.
Brief Title: ReAL Trial (Rectal Anastomotic seaL)
Acronym: ReAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 131/2019
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-05

CONDITIONS: Rectal Cancer
Keywords: colorectal anastomosis; leakage
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyanoacrylate (Experimental): the anastomotic reinforcement with nebulized cyanoacrylate glue using the special short catheter device for open surgery or the laparoscopic catheter.
  Interventions: Procedure: Cyanoacrylate reinforcement
- No reinforcement (Active Comparator): No reinforcement will be applied on the anastomosis line
  Interventions: Procedure: No reinforcement

INTERVENTIONS:
Procedure: Cyanoacrylate reinforcement — Anastomosis Reinforcement with with nebulization of 1cc of glue on the anastomosis line
  Arms: Cyanoacrylate
Procedure: No reinforcement — Nothing applied on the anastomosis line
  Arms: No reinforcement

SUMMARY:
The problem of anastomotic leak is particularly relevant in rectal surgery. Many risk factors have been recognized in the onset of this complication. Preventing the anastomotic leak can bring benefits to the patient and the health system.

Several attempts have been proposed to reduce the risk of anastomotic leakage in rectal cancer surgery including suture protection with omental flap and external suture reinforcement by biological glue or mesh.

Cyanoacrylate (Glubran 2®) is a synthetic glue with sealing, adhesive and hemostatic properties widely used in surgery. The sealing effect creates an antiseptic barrier against bacteria.

The hypothesis is that the application of nebulized cyanoacrylate to the colo-rectal anastomosis in open or laparoscopic/robotic rectal surgery can prevent the leakage

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most common cause of cancer-related death in male and the third in females in Western Countries accounting for more than 500,000 deaths in 2013 worldwide.

One of the most worrying postoperative complication in colorectal surgery is the anastomotic leak which can occur in about 10-15% of the cases.

This complication severely impact clinical outcomes with increased risk of death or permanent stoma, higher risk of local recurrence) and relevant increase in hospital costs (length of hospital stay, admission to intensive care, re-interventions).

The problem of anastomotic leak is particularly relevant in rectal surgery. The more distal the anastomosis, the higher the likelihood of failure, with resection of a distal rectal cancer having almost a five-fold increased risk of anastomotic leak compared with resection for colon cancer.

In fact, anastomotic Leakage (AL) is the most severe complication after Low anterior resection of rectum for cancer, occurring between 3 and 24 % of patients.

Many risk factors have been recognized in the onset of this complication, including gender (male patient have a higher anastomotic leak rate), malnutrition, obesity an diabet, american society anesthesiologists (ASA) score, tobacco use, cardiovascular disease, immunosuppression, use of NSAID, preoperative pelvis radiation.

Other intraoperative risk factors considered are the splenic flexure mobilization with proximal ligation of the inferior mesenteric artery (IMA), positive intraoperative Air-Leak Test and the perfusion of the anastomosis.

Temporary fecal diversion has also been suggested (although a diverting stoma mitigates the clinical consequences of an anastomotic leak but does not prevent it.

Other intraoperative technical factors include the use of single or double stapled anastomotic techniques, with or without transanal reinforcing sutures.

Therefore, preventing the anastomotic leak can bring benefits to the patient and the health system.

All the risk factors described above represent the rationale that justifies the use of intraoperative procedures to prevent the anastomotic leak, such as additional manual stiches to the mechanical suture and / or patches of collagen (proper reinforcement or buttressing) or of sealants.

Several attempts have been proposed to reduce the risk of AL in rectal cancer surgery including suture protection with omental flap and external suture reinforcement by biological glue or mesh.

Some Authors have reported good results of reinforcement of the colon anastomosis with cyanoacrylate glue. in a porcine model.

Cyanoacrylate is a synthetic glue with sealing, adhesive and haemostatic properties widely used in surgery. Furthermore the sealing effect creates an antiseptic barrier against bacteria.

Several clinical studies have described the utility of cyanoacrylate glue mainly in vascular surgery, urology and bariatric surgery.

Considering its mechanical, physical, biological properties and its safety, cyanoacrylate glue could facilitate the healing of the colorectal anastomosis reducing leak rate, without negative effects on perfusion.

The hypothesis is that the application of nebulized cyanoacrylate to the colo-rectal anastomosis in open or laparoscopic/robotic rectal surgery can prevent the leakage

ELIGIBILITY:
Inclusion Criteria:

* Resectable, histologically proven primary adenocarcinoma of the High-medium rectum without internal and/or external sphincter muscle involvement.
* Distal margin of the tumor at least 8 cm form the anal verge
* Staged as follows prior to neoadjuvant chemoradiation: Stage T2 - T4 at MRI
* Patient classified T3-T4 will undergo neoadjuvant chemoradiation if the cancer is located in the extraperitoneal rectum

Exclusion Criteria:

* Squamous cell carcinoma
* Adenocarcinoma Stage T1,
* T4 with one of the following: with pelvic side wall involvement, requiring sacrectomy, requiring prostatectomy (partial or total)
* Unresectable primary rectal cancer or Inability to complete R0 resection.
* Rectal cancer under 8 cm from the anal verge requiring colo-anal or ultra low rectal anastomosis
* Recurrent rectal cancer
* Previous pelvic malignancy
* Inability to sign the informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-12-02 (Estimated); Study Completion 2021-07-02 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak | 30 days
  leakage of the colorectal anastomosis clinically proven or with two sides X-ray

SECONDARY OUTCOMES:
length of hospital stay | 30 days
  duration of hospital stay
Blood loss | 1 day
  the amount of bleeding during the operation
Surgical site infection | 30 days
  purulent discharge from the wound with positive culture
Postoperative complications | 30 days
  complications after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Donato Altomare, Prof, Principal Investigator — Societa Italiana di Chirurgia ColoRettale; Arcangelo Picciariello, MD, Principal Investigator — Societa Italiana di Chirurgia ColoRettale
Locations (1):
- Dept of Emergency and Organ transplantation - University of Bari, Bari, Italy

REFERENCES:
- [Result] Thomas MS, Margolin DA. Management of Colorectal Anastomotic Leak. Clin Colon Rectal Surg. 2016 Jun;29(2):138-44. doi: 10.1055/s-0036-1580630. PMID 27247539
- [Result] de la Portilla F, Zbar AP, Rada R, Vega J, Cisneros N, Maldonado VH, Utrera A, Espinosa E. Bioabsorbable staple-line reinforcement to reduce staple-line bleeding in the transection of mesenteric vessels during laparoscopic colorectal resection: a pilot study. Tech Coloproctol. 2006 Dec;10(4):335-8. doi: 10.1007/s10151-006-0303-0. Epub 2006 Nov 27. PMID 17115313
- [Result] Wiggins T, Markar SR, Arya S, Hanna GB. Anastomotic reinforcement with omentoplasty following gastrointestinal anastomosis: A systematic review and meta-analysis. Surg Oncol. 2015 Sep;24(3):181-6. doi: 10.1016/j.suronc.2015.06.011. Epub 2015 Jun 17. PMID 26116395
- [Result] Boersema GSA, Vennix S, Wu Z, Te Lintel Hekkert M, Duncker DGM, Lam KH, Menon AG, Kleinrensink GJ, Lange JF. Reinforcement of the colon anastomosis with cyanoacrylate glue: a porcine model. J Surg Res. 2017 Sep;217:84-91. doi: 10.1016/j.jss.2017.05.001. Epub 2017 May 10. PMID 28595813
- [Result] Montanaro L, Arciola CR, Cenni E, Ciapetti G, Savioli F, Filippini F, Barsanti LA. Cytotoxicity, blood compatibility and antimicrobial activity of two cyanoacrylate glues for surgical use. Biomaterials. 2001 Jan;22(1):59-66. doi: 10.1016/s0142-9612(00)00163-0. PMID 11085384
- [Result] Wu Z, Boersema GS, Vakalopoulos KA, Daams F, Sparreboom CL, Kleinrensink GJ, Jeekel J, Lange JF. Critical analysis of cyanoacrylate in intestinal and colorectal anastomosis. J Biomed Mater Res B Appl Biomater. 2014 Apr;102(3):635-42. doi: 10.1002/jbm.b.33039. Epub 2013 Oct 24. PMID 24155114
- [Derived] Tomasicchio G, Martines G, Tartaglia N, Buonfantino M, Restini E, Carlucci B, Giove C, Dezi A, Ranieri C, Logrieco G, Vincenti L, Ambrosi A, Altomare DF, De Fazio M, Picciariello A. Suture reinforcement using a modified cyanoacrylate glue to prevent anastomotic leak in colorectal surgery: a prospective multicentre randomized trial : The Rectal Anastomotic seaL (ReAL) trial. Tech Coloproctol. 2024 Aug 5;28(1):95. doi: 10.1007/s10151-024-02967-7. PMID 39103661

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT03941938/Prot_SAP_001.pdf